CLINICAL TRIAL: NCT05712239
Title: Effect of Adding Lumbar Core Stability Exercises to Cervical and Scapular Stabilization Exercises and Advices on Chronic Non- Specific Neck Pain
Brief Title: Effect of Lumber Core Stability Exercises on Chronic Non-specific Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hend Wageh, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003950
Record Dates: First submitted 2023-01-26; First posted 2023-02-03 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: To confirm blindness, all patients will be unaware of the group allocation and the exercises performed by the other group. Also, the pictures of craniovertebral angle will be coded before being measured
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Advices Group (Other): Patients in this group will take only advices about their postures and activities of daily living
  Interventions: Other: Advices
- Cervical and scapular stabilization Group (Active Comparator): Patients in this group will take advices and stability exercises for neck and scapula
  Interventions: Other: Advices; Other: Cervical and Scapular Stabilization Exercises
- Neck, scapular and lumber stabilization Group (Experimental): Patients in this group will take advices, and stability exercises for neck, scapula and lumber spine
  Interventions: Other: Advices; Other: Cervical and Scapular Stabilization Exercises; Other: Lumber Core Stability Program

INTERVENTIONS:
Other: Advices — The advices will include patient's reassurance and description of possible causes of neck pain such as poor working ergonomics, common bad postures especially while using electronic devices for long periods and not adjustable sleeping pillows. Also, patient will be educated how to modify these different causes and asked to apply gentle neck range of motion exercises
Other: Cervical and Scapular Stabilization Exercises — Deep neck flexor training will be performed in neurodevelopment stages (supine at first week using pressure biofeedback unit , prone at second week, quadrupedal at third week, bipedal at fourth week).
  Scapular stabilization exercises will include modified prone cobra, trapezius muscle exercise progression (3 stages), wall press and extension of the thoracic spine using foam roller. The modified prone cobra and the first stage of trapezius muscle exercise progression will be applied during the first two weeks. The second and third stages of trapezius muscle exercise will be applied during the last two weeks of our rehabilitation program. All exercises will be applied for 10 repetitions with 6-10 sec hold for 3 sets with 20 sec rest between each set. While wall press and thoracic extension exercises will be applied throughout the 4 weeks for 3 sets of 10 repetitions with 20 sec rest between each set.
  Arms: Cervical and scapular stabilization Group; Neck, scapular and lumber stabilization Group
Other: Lumber Core Stability Program — The program will be performed in three stages: activation, dynamic stabilization, and advanced core strengthening stages. Each stage will be applied for 4 sessions.
  The activation stage will be based on the learning to activate transversus abdominis muscle from crock lying position using pressure biofeedback unit. In the dynamic stabilization stage, the patient will be instructed to slowly raise both arms in the scapular plan then return to the sides while maintaining the transversus abdominis muscle activation. Also, the patient will apply bridging exercise in this stage. The advanced core strengthening stage will include prone plank and side plank (right and left sides). All the exercises will be applied for 10 repetitions with 6-10 sec hold for 3 sets. The rest of 20 sec will be taken between each set.
  Arms: Neck, scapular and lumber stabilization Group

SUMMARY:
Chronic non-specific neck pain patients will be enrolled in 3 groups in this study including passive, active control and experimental groups to determine the effect of adding lumbar core stability exercises to patient's advices and cervical and scapular stabilization exercises. For the last two groups, the sessions will be applied 3 times per week for 4 weeks. All the outcomes will be measured after patient's enrollment and at the end of 4 weeks to determine the difference between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent cervical pain for more than 12 weeks without specific diagnosis (chronic non-specific neck pain).
* BMI less than 30 kg/m2.
* Pain intensity on VAS should be more than 3.
* Patient will be able and motivated in completing the study.
* Psychologically & mentally stable.

Exclusion Criteria:

* Red Flag's symptoms including a history of major trauma, persistent night pain, bladder or bowel dysfunction, and/or lower or upper extremity neurological deficit.
* Pregnant women.
* Recent or old fractures at spine or upper limbs.
* Congenital, or acquired postural deformity.
* No previous neck or spinal or shoulder surgery.
* No current pathologies (e.g. Disc lesion, nerve root compression, canal stenosis, spinal tumor, spinal infection, systemic inflammatory diseases, …).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-02-05 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
change in pain intensity | This outcome will be assessed at the first day and after 4 weeks following end of treatment
  Pain intensity will be assessed by using Visual analogue scale (VAS). It is horizontal line with 10 cm length, with Zero marked at one end representing no pain and 10 marked at the other end representing worst imaginable pain.
change in functional disability | This outcome will be assessed at the first day and after 4 weeks following end of treatment
  Functional disability will be assessed using Arabic version of neck disability index. The patients will be asked to make a mark in each section which most closely described their problem. Each section consists of six potential responses for each item ranging from no disability (0) to total disability (5). Thus, The NDI score ranges between 0-100, with higher scores indicating greater perceived disability. The score of less than 4 indicates no disability, 5-14 mild disability, 15-24 moderate disability, 25-34 severe disability, and scores greater than 35 complete disabilities.

SECONDARY OUTCOMES:
change in Craniovertebral angle degree (CVA) | This outcome will be assessed at the first day and after 4 weeks following end of treatment
  To measure CVA, the patient will be captured from the left side after putting landmarks on seventh cervical vertebra (c7) and tragus of the ear. The photograph will be taken and analyzed with kinovea software by drawing a horizontal line passing through C7 and line connecting between the tragus of the ear and C7 and measuring the angle between these lines. As the value of CVA decreases, the degree of FHP increases
change of of deep neck flexor muscles (DNF) activation | This outcome will be assessed at the first day and after 4 weeks following end of treatment
  DNF activation will be assessed by Craniocervical flexion test using Pressure biofeedback unit
change of deep neck flexor (DNF) endurance | This outcome will be assessed at the first day and after 4 weeks following end of treatment
  DNF endurance will be assessed by Neck flexor endurance test
change of trunk flexor muscle endurance | This outcome will be assessed at the first day and after 4 weeks following end of treatment
  Trunk flexor muscle endurance will be assessed by Trunk flexion test (McGill's test)
change of trunk extensor muscle endurance | This outcome will be assessed at the first day and after 4 weeks following end of treatment
  Trunk extensor muscle endurance will be assessed by Trunk extension test (Sorenson Test)
change of lateral trunk muscle endurance | This outcome will be assessed at the first day and after 4 weeks following end of treatment
  Lateral trunk muscle endurance will be assessed Side plank test for left and right sides

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Egypt